CLINICAL TRIAL: NCT01265225
Title: Prognostic Value of Stem Cell Related Markers CD24, CD44, CD326 and EPCR, for Predicting Breast Cancer Recurrence in Tumor Stages 0-II
Brief Title: Prognostic Value of Stem Cell Related Markers
Status: Withdrawn | Type: Observational
Why Stopped: no finance
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Dr. I. Schnirer, Baruch Padeh Poriya Medical Center
Other Study IDs: 10.CTIL
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: breast cancer stages 0-II
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of the investigators study is to identify a prognostic marker that will evaluate the probability of recurrence in patients with stage 0-II breast cancer following surgery to remove the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Ductal Carcinoma in Situ
* DCIS + Microinvasion stages 1 or 11 without positive lymph nodes

Exclusion Criteria:

* tumor specimen with higher than grade II
* BRACA 1 or BRACA 2 mutation
* Neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 tumor specimens from women with grade 0-11 ductal breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Baruch PMC, Poria – Neve Oved, Lower Galilee, Israel